CLINICAL TRIAL: NCT02714231
Title: A Randomized Controlled Trial of 2 Different Methods for Pain Relief During Intrauterine Device Insertion
Brief Title: Oral Diclofenac Sodium Versus Oral Hyoscine Butyl Bromide During Intrauterine Device Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DS-HB
Record Dates: First submitted 2016-03-14; First posted 2016-03-21 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Family Planning
MeSH Terms: interventions — Diclofenac; Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diclofenac (Experimental): oral diclofuhenac sodium
  Interventions: Drug: diclofenac sodium (cataflam)
- hyoscine (Active Comparator): oral hyoscine butyl bromide
  Interventions: Drug: hyoscine butyl bromide (buscopan)

INTERVENTIONS:
Drug: diclofenac sodium (cataflam) — The patients in the study group will take one tablet of cataflam 50 mg 30 min before the scheduled time of the procedure
  Arms: diclofenac
Drug: hyoscine butyl bromide (buscopan) — The patients in the study group will take one tablet of buscopan 10 mg 30 min before the scheduled time of the procedure
  Arms: hyoscine

SUMMARY:
The aim of our study is to compare the analgesic effect of oral diclofenac sodium versus oral hyoscine butyl bromide during intrauterine device insertion.

ELIGIBILITY:
Inclusion Criteria:

* Women not taken analgesics or anxiolytics in the 24 hours prior insertion
* Women not taken misoprostol prior to intrauterine device insertion
* Women who will accept to participate in the study

Exclusion Criteria:

* Any contraindication to intrauterine device placement

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Mean pain score during insertion | intraoperative

SECONDARY OUTCOMES:
Patient satisfaction score | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: ahmed abbas, MD, Principal Investigator — Woman health hospital Assiut
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes